CLINICAL TRIAL: NCT02874716
Title: An Impact Evaluation of the Private Provider Interface Agency Program on Quality of Tuberculosis Care: A Standardized Patient Study in Patna, India
Brief Title: Quality of Tuberculosis Care in Urban Patna, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: World Bank (Other); Institute of Socio-Economic Research on Development and Democracy (ISERDD) (Unknown); ACCESS Health International (Other)
Responsible Party: Principal Investigator, Madhukar Pai, Canada Research Chair in Epidemiology & Global Health, Director of McGill Global Health Programs, Associate Director of McGill International Tuberculosis Centre, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: OPP1091843-1
Record Dates: First submitted 2016-08-07; First posted 2016-08-22 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Tuberculosis
Keywords: Quality of Care; Standardized Patients
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tuberculosis Program (PPIA) (Experimental): In Patna, 171 of the 321 participants were randomly selected to be sensitized and engaged into the program in Phase 1, and subsequently to receive the benefits of the PPIA intervention. Providers in the PPIA arm if engaged into the program will receive the benefits of the program, including but not limited to: ability to provide presumptive TB patients and TB cases vouchers for free or subsidized diagnostic testing and free first line anti-TB treatment (TB cases only); reimbursements for subsidized tests and anti-TB treatment; financial incentives to providers based on certain indicators; training opportunities, and access to a referral network.
  Interventions: Other: Tuberculosis Program (PPIA)
- No Tuberculosis Program (Non-PPIA) (No Intervention): The remaining part of the sample in Patna selected randomly will be phased into the program at least a year after the PPIA arm in Phase 2. However, during the year of the study, they will not be engaged into the program.

INTERVENTIONS:
Other: Tuberculosis Program (PPIA) — The intervention includes a variety of (1) non-financial incentives that are intended to reduce clinical and financial costs for presumptive TB patients and TB cases for diagnostic testing and treatment (free sputum microscopy, free digital chest X-ray, free or subsidized drug-susceptibility testing (DST), free first line anti-TB treatment), (2) training or certified medical education sessions for the providers from the PPIA, and (3) financial incentives to engaged providers for patient registration, diagnostic testing, treatment initiation, and treatment adherence. Meanwhile, health camps, advertising, and other advocacy efforts are aimed to raise awareness in the communities.
  Other Names: Private Provider Interface Agency Program
  Arms: Tuberculosis Program (PPIA)

SUMMARY:
The purpose of this study is to evaluate the impact of the Private Provider Interface Agency (PPIA) program on quality of health care. The PPIA is a tuberculosis pilot program implemented in the private health sector of urban Patna in the state of Bihar, India.

DETAILED DESCRIPTION:
By taking advantage of a randomized roll-out design of the PPIA program in urban Patna, this evaluation aims to determine the causal effects of the program on quality of health care among private sector health providers. The evaluation is embedded in an existing quality of care surveillance project that uses standardized patients to assess the quality of tuberculosis (TB) care in urban Patna. Below is a description of (1) the TB intervention implemented by the PPIA, (2) the quality of TB care (QuTUB) surveillance project, and (3) the randomized roll-out of the PPIA program among a subset of providers in order to isolate the impact of the program on quality of care.

The entire program and its implementation are external to the researchers. To better understand the impact of the program using an already approved design, the researchers use a stepped-wedge design that involves a sequential roll out of the program to a subset of providers over a period of time where the order of roll-out is randomized.

1. PPIA intervention: Between January 2014 and December 2016, the pilot PPIA program was independently implemented by the non-governmental organization World Health Partners (WHP) in urban Patna. In its role as the PPIA in Patna, WHP's aim is to strengthen existing efforts to control TB through engagement of the private health sector. Through this network, the objectives are to facilitate early and accurate diagnosis with proper notification of cases and to ensure appropriate treatment and treatment adherence to completion among TB patients in the private sector. This is done by establishing a network and engaging four types of private health sector actors who are of vital importance for TB advocacy and treatment efforts: (i) formal providers, who are qualified doctors at hospitals, nursing homes, or outpatient clinics who receive presumptive TB cases or treat TB cases, (ii) informal providers, who are non-allopathic providers or less than fully qualified practitioners, including practitioners of alternative medicines Ayurveda, Yoga and Naturopathy, Unani, Siddha, and Homeopathy and other practitioners with minimum or no qualifications, (iii) chemists/pharmacists with a drug license, medicine stock, and anti-TB drugs for sale, and (iv) diagnostic laboratories that conduct sputum smear microscopy and/or chest X-rays, and GeneXpert drug susceptibility testing. The pilot will serve as a model for private health sector involvement in national TB control and will be used to inform similar programs in other urban Indian settings.
2. Quality of care surveillance: The QuTUB project is a part of the PPIA monitoring efforts and runs in parallel to the program scale up and expansion. The objective of the QuTUB project is to capture levels of quality of care through standardized patients ("mystery shoppers" or "fake patients"), who are individuals recruited locally and trained to portray four different TB cases. Developed by a Technical Advisory Group and benchmarked against the Standards of TB Care of India, the cases were designed to reflect different stages of TB disease progression, some with previous interactions with the health system upon presentation to a health care provider. Outcomes captured by the standardized patients through an exit questionnaire given to them within 2 hours of their interaction with providers include: history questions asked by the provider, laboratory tests ordered, medicines dispensed or prescribed, and referrals made.
3. Randomized roll-out evaluation approach: In December 2014, WHP was interested in trying to further understand the causal impact of their program on diagnostic processes, and there was an opportunity to remove the selection bias and attribute differences in quality of care solely to the program by taking advantage of a randomized roll-out expansion plan of the PPIA program among a subset of providers. In collaboration with the PPIA Patna team, this study takes an intention-to-treat and instrumental variables evaluation approach through selective enrollment of a subset of providers in the second round of program scale-up across urban Patna. The researchers note that the subset of providers are those who were not purposively selected in the earlier round of enrollment and therefore may be those who see fewer TB patients, or those who were reluctant to enroll into the program during the first rounds of program expansion. Therefore, the impact of the program on this group may be different from among those who were enrolled previously. Under this approach, it was agreed that for the evaluation eligible formal providers would be engaged. For this, the researchers provided WHP with a list of 321 randomly selected providers among those who were not already enrolled at the beginning of 2015. Providers on this list were randomly allocated to two groups: one group (treatment) of 171 eligible formal providers would be sensitized and engaged, and the other group (control) of 150 eligible formal providers would not be engaged until the QuTUB study team is able to complete end-line data collection in 2016, after a year or more. Selection into program roll-out groups was randomized. The study group includes formal providers who would see a pulmonary TB case and self-reported low caseloads. Standardized patients are sent to both groups before any intervention for baseline measures of quality of care, and the standardized patients would return again before the control group begins to receive the intervention for an end-line measure. The entire intervention in Patna is implemented by the PPIA and is separate from the research team implementing the quality of care surveillance and evaluation. Care is taken to ensure that the evaluation team will be in the field independently of the implementation.

Analysis:

Intention-to-treat analysis and instrumental variables will be conducted after determining (i) that the treatment assignment can serve as a good instrument by: a strong correlation to the actual enrollment statuses of the providers regardless of treatment assignment, being uncorrelated with the outcomes, and only being connected to the outcomes through actual enrollment in the program, and (ii) balance at baseline between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Formal providers (with Bachelor of Medicine, Bachelor of Surgery (MBBS) degree and higher) who were not enrolled in the urban PPIA program as of January 2015
* Daily outpatients of 20 or fewer (self-reported)

Exclusion Criteria:

* Formal providers enrolled in the urban PPIA program as of January 2015
* Formal providers who do not see adult pulmonary patients (e.g., pediatricians, orthopedists)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Correct case management | one year
  Correct case management is defined as the proportion of interactions (across all standardized patient (SP) cases) or proportion of providers (by SP case) in which providers managed the case according to the Standards for Tuberculosis Care in India (STCI) within the PPIA program vs. outside the PPIA. Depending on the SP case, the outcome is an index composed of actions a provider did during the interaction with the SP: correct diagnostic tests ordered, correct or harmful treatment prescribed, or referral to a qualified health care provider. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.

SECONDARY OUTCOMES:
Essential history checklist | one year
  Essential history checklist is defined as the average proportion of essential history questions asked by the practitioner during an interaction for tuberculosis benchmarked against the Standards of Tuberculosis Care in India guidelines. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Referral for further management | one year
  Referral for further management is defined as the proportion of interactions in which the provider refers the simulated patient to a qualified provider or another facility and the name, if specified to the SP. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Suspicion of tuberculosis | one year
  Suspicion of tuberculosis is defined as the proportion of interactions in which the provider mentions tuberculosis or states that the simulated patient has tuberculosis. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Initiation of TB treatment | one year
  Initiation of TB treatment is defined as the proportion of interactions in which the provider initiates the simulated patient on TB treatment. After each interaction, the SP purchases any medicines ordered by the provider. These details are collected on an exit questionnaire; active ingredients are investigated; and medicines are coded separately by two clinicians on the research team.
Number of lab tests ordered | one year
  Number of lab tests ordered is defined as the average number of lab tests ordered per interaction by providers. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Lab tests ordered | one year
  Lab tests ordered is defined as the proportion of interactions in which the provider orders specific TB diagnostic tests (e.g. chest X-ray, sputum acid-fast bacillus (AFB) testing, GeneXpert) or other types of tests for the simulated patient. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Number of medicines | one year
  Number of medicines is defined as the average number of medicines ordered per interaction. After each interaction, the SP purchases any medicines ordered by the provider. These details are collected on an exit questionnaire; active ingredients are investigated; and medicines are coded and categorized by two clinicians on the research team.
Medicine type | one year
  Medicine type is defined as the types of medicines ordered (e.g., antibiotics, steroids, fluoroquinolones, and others) during the simulated patient interactions. After each interaction, the SP purchases any medicines ordered by the provider. These details are collected on an exit questionnaire; active ingredients are investigated; and medicines are coded and categorized by two clinicians on the research team.
Rates of case registration for practitioners networked in the program | one year
  Rates of case registration is defined as the proportion of interactions in which providers who are networked in the PPIA program registers the simulated patient into the program. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Vouchers received | one year
  Vouchers received is defined as the proportion of PPIA vouchers or referral coupons given to the simulated patient for any of the actions that could have resulted in a voucher or referral coupon only among providers who are in the PPIA program. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Patient costs | one year
  Patient costs is defined as the average amount charged to the simulated patients by providers per interaction for the entire visit. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.
Consultation, medicine, and test costs to patients | one year
  The outcome for consultation, medicine, and test costs to patients is defined as the average amount charged for consultation, medicines, and tests (if itemized) by providers per interaction. These details are extracted from an exit questionnaire that is completed by the SP within 2 hours of the interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Pai, MD, PhD, Principal Investigator — McGill University; Jishnu Das, PhD, Principal Investigator — World Bank

REFERENCES:
- [Background] Das J, Kwan A, Daniels B, Satyanarayana S, Subbaraman R, Bergkvist S, Das RK, Das V, Pai M. Use of standardised patients to assess quality of tuberculosis care: a pilot, cross-sectional study. Lancet Infect Dis. 2015 Nov;15(11):1305-13. doi: 10.1016/S1473-3099(15)00077-8. Epub 2015 Aug 9. PMID 26268690